CLINICAL TRIAL: NCT04416217
Title: Adrenal Suppression in Pediatric Eosinophilic Esophagitis Treated With Topical Steroids - A Multicenter, Prospective, Observational Safety Study
Brief Title: Eosinophilic Esophagitis Steroid Safety Study
Acronym: EESY
Status: Completed | Type: Observational
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Noam Zevit, Attending Pediatric Gastroenterologist, Schneider Children's Medical Center, Israel
Other Study IDs: 0521-19-RMC
Record Dates: First submitted 2020-05-24; First posted 2020-06-04 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Eosinophilic Esophagitis
Keywords: Steroid , bone mineral density , DEXA , Adrenal
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Topical Steroid Treatment: Pediatric patients with eosinophilic esophagitis scheduled to begin topical steroid treatment for the treatment of their condition. The type of topical steroid is not limited and is at the discretion of the treating physician as are dosing and concomitant treatments.

SUMMARY:
This observational study will follow pediatric patients with eosinophilic esophagitis who are scheduled to begin topical steroid treatment, from the initiation of treatment longitudinally to determine the safety profile of the drug.

ELIGIBILITY:
Inclusion Criteria:

1. Age <18 years at the time of enrollment.
2. Males and Females are included.
3. Patients diagnosed with EoE as defined by age appropriate signs of esophageal dysfunction (in older children and adolescents - dysphagia, impacted food bolus, foreign body impaction, vomiting, and GERD not responsive to high dose proton pump inhibitors. In infants and young children - failure to thrive, poor feeding, vomiting, food bolus impaction)
4. Histopathological finding of ≥15 eosinophils/high power field (X400) on at least one esophageal biopsy.
5. After discussing the available treatment options with the gastroenterologist, the patient has chosen oral topical steroid treatment (either as a first treatment or after failure of other dietary or medical treatment).

Exclusion Criteria:

1. Known alternative causes of esophageal eosinophilia.
2. Legal guardian unable or unwilling to sign informed consent..
3. Known allergy to topical steroids ingredients
4. Patient will not be available for follow-up for at least the 3 month assessment and ACTH test.
5. Known pregnancy
6. Use of oral systemic steroids in the 6 months prior to inclusion in the study. Use of systemic steroids once in the study will not lead to study termination, but such use will need to be reported in the medication changes and use page of the following visit.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients diagnosed with eosinophilic esophagitis for whom following discussion between the patient/gaurdians and physician treatment with topical steroids are planned.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Adrenal suppression | 3 months
  Rates of pathological adrenocorticotropic hormone (ACTH) tests at 3 and 12 months of topical steroid use
Adrenal suppression | 12 months
  Rates of pathological adrenocorticotropic hormone (ACTH) tests at 3 and 12 months of topical steroid use
Growth failure | 12 months
  Rates of decreased Height for age after 12 months of treatment.
Growth failure | 36 months
  Rates of decreased Height for age after 12 months of treatment.

SECONDARY OUTCOMES:
Bone mineral density | 12 months
  Decrease in bone mineral density between first and second dual energy x-ray absorptiometry (DEXA)
Bone mineral density | 3 years
  Decrease in bone mineral density between first and second dual energy x-ray absorptiometry (DEXA)
Hyperglycemia | 3 months
  Rates of elevated fasting glucose after 3 and 12 months of treatment
Hyperglycemia | 12 months
  Rates of elevated fasting glucose after 3 and 12 months of treatment
Elevated Liver Enzymes | 3 months
  Elevated ALT
Histological remission 3 months | 3 months
  Histological remission at endoscopy timepoints
Histological remission 12 months | 12 months
  Histological remission at endoscopy timepoints
Clinical remission | 3 months
  Clinical remission at endoscopy time points according to PEESS v.2
Clinical remission | 12 months
  Clinical remission at endoscopy time points according to PEESS v.2

CONTACTS AND LOCATIONS:
Locations (4):
- Athens Children's Hospital "AGIA SOPHIA", Athens, Greece
- Institute of Gastroenterology, Nutrition and Liver Diseases; Schneider Children's Medical Center of Israel, Petah Tikva, Israel
- Italy (2):
  - Department of Woman, Child and General and Specialized Surgery, University of the Campania "Luigi Vanvitelli", Naples
  - Maternal and Child Health Department, Sapienza, Rome

REFERENCES:
- [Background] Armstrong DH. Portable sampler for microorganisms in incinerator stack emissions. Appl Microbiol. 1970 Jan;19(1):204-5. doi: 10.1128/am.19.1.204-205.1970. PMID 5415218
- [Background] Hsu S, Wood C, Pan Z, Rahat H, Zeitler P, Fleischer D, Menard-Katcher C, Furuta GT, Atkins D. Adrenal Insufficiency in Pediatric Eosinophilic Esophagitis Patients Treated with Swallowed Topical Steroids. Pediatr Allergy Immunol Pulmonol. 2017 Sep 1;30(3):135-140. doi: 10.1089/ped.2017.0779. PMID 29062584
- [Background] Golekoh MC, Hornung LN, Mukkada VA, Khoury JC, Putnam PE, Backeljauw PF. Adrenal Insufficiency after Chronic Swallowed Glucocorticoid Therapy for Eosinophilic Esophagitis. J Pediatr. 2016 Mar;170:240-5. doi: 10.1016/j.jpeds.2015.11.026. Epub 2015 Dec 11. PMID 26687577
- [Background] Harel S, Hursh BE, Chan ES, Avinashi V, Panagiotopoulos C. Adrenal insufficiency exists for both swallowed budesonide and fluticasone propionate in the treatment of eosinophilic esophagitis. J Pediatr. 2016 Jul;174:281. doi: 10.1016/j.jpeds.2016.02.056. Epub 2016 Mar 19. No abstract available. PMID 27004676
- [Background] Philpott H, Dougherty MK, Reed CC, Caldwell M, Kirk D, Torpy DJ, Dellon ES. Systematic review: adrenal insufficiency secondary to swallowed topical corticosteroids in eosinophilic oesophagitis. Aliment Pharmacol Ther. 2018 Apr;47(8):1071-1078. doi: 10.1111/apt.14573. Epub 2018 Mar 5. PMID 29508432